CLINICAL TRIAL: NCT06648889
Title: A Multicenter, Single-arm Phase II Study to Assess the Safety, Tolerability, and Efficacy of Isatuximab in Adult Patients With Cytologic or Molecular Relapsed/Refractory CD38 Positive T-cell Acute Lymphoblastic Leukemia (GMALL-Isatuximab)
Brief Title: Isatuximab in Adult Patients With Cytologic or Molecular Relapsed/Refractory CD38 Positive T-cell Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Nicola Goekbuget, Dr. Nicola Gökbuget, Head of Trial Center, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMALL-Isatuximab; 2023-507899-47-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-15; First posted 2024-10-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: T-ALL
Keywords: R/R or MRD CD38-positive T-ALL
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — isatuximab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GMALL-Isatuximab (Experimental): Cohort 1: In this Cohort, Isatuximab shall be implemented as part of a combination therapy for patients with R/R T-ALL, defined as bone marrow infiltration of ≥5% (R/R T-ALL).
  Cohort 2: In this Cohort, Isatuximab shall be implemented as single drug treatment for patients with molecular failure/relapse. Cohort 2 will include patients with hematologic remission (bone marrow blast count <5%) of T-cell ALL, but with molecular failure or molecular relapse (MRD+ T-ALL).
  Interventions: Drug: Isatuximab

INTERVENTIONS:
Drug: Isatuximab — Cohort 1: All patients will receive two cycles of induction therapy with standard chemotherapy, Bortezomib and Isatuximab. Isatuximab maintenance may be administered in patients with CR until SCT, progression/relapse, unacceptable toxicity, physicians' decision to change treatment or withdrawal of consent.
  Other Names: Bortezomib
Drug: Isatuximab — Cohort 2: All patients will receive at least one cycle with Isatuximab. Each cycle will be 4 weeks in duration. Isatuximab will be administered until SCT, hematologic relapse including extramedullary, unacceptable toxicity, physicians' decision, or withdrawal of consent.

SUMMARY:
The planned trial offers treatment cohorts for patients with full cytologic relapse (R/R ALL - Cohort 1), as well as for patients with molecular failure/relapse (MRD+ ALL - Cohort 2). Basically, the study aims to develop data for optimization of first-line therapy of T-ALL, either by modification of standard induction with Isatuximab or by establishing a post-induction therapy for eradication of MRD and thereby evaluates in parallel two different strategies.

ELIGIBILITY:
Inclusion Criteria:

- Patients with CD38 positive T-ALL fitting either to the definitions for cohort 1 or cohort 2:

Cohort 1: In relapse or with primary refractory disease defined as ≥5% blasts in bone marrow after at least three chemotherapy cycles (induction I-II, consolidation I) with the following additional specifications:

* early relapse within 12 months from first achievement of CR or
* late relapse later than 12 months from first achievement of CR or
* primary refractory disease without any CR or
* any relapse after stem cell transplantation or
* any refractory relapse, defined as no response to at least one salvage therapy or
* any second or later relapse and
* Availability of patient material with blast cells (bone marrow or peripheral blood) for central MRD assessment or availability of respective predefined marker.

Cohort 2: In complete hematological remission (defined as less than 5% blasts in bone marrow and no evidence of extramedullary disease) after at least three chemotherapy cycles (induction I-II, consolidation I)

* Detection of quantifiable MRD at a level of ≥10-4, either as molecular failure without prior achievement of molecular remission or molecular relapse after prior achievement of molecular remission
* MRD assay at the central reference lab with at least one marker a minimum sensitivity of 10-4
* MRD detection for study inclusion after an interval of at least 2 weeks from last systemic chemotherapy including antibody therapy
* (in patients without clonal molecular MRD marker, MRD testing can be based on flow-cytometry established in reference laboratory)

ECOG status:

* Cohort 1: 0-2
* Cohort 2: 0-1

Age ≥ 18 years Evidence of a personally signed and dated informed consent indicating that the patient has been informed of all pertinent aspects of the study Patient must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Regeneration from last chemotherapy defined as follows:

Cohort 1:

* Platelets ≥10.000/uL (platelet transfusion allowed)
* Hemoglobin ≥ 7.5 g/dl (red blood cell transfusion allowed)

Cohort 2:

* Neutrophils ≥1.000/uL
* Platelets ≥50.000/uL
* Hemoglobin ≥9 g/dl

Adequate liver function defined as follows:

* Bilirubin ≤ 1.5 ULN (unless Gilbert Meulengracht disease or classified as result of liver infiltration by investigator)
* AST and ALT ≤ 2.5 x ULN (unless classified as result of liver infiltration by investigator)

Adequate renal function defined as follows:

* Serum creatinine ≤ 2 x ULN
* Any serum creatinine level associated with a calculated creatinine clearance ≤ 40 mL/min
* Negative pregnancy test in women of childbearing potential (WOCBP)
* WOCBP must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously.
* Men who are sexually active with a WOCBP must agree to use a barrier method of contraception
* Participation in the registry of the German Multicenter Study Group for Adult ALL (GMALL)

Exclusion Criteria:

* Extramedullary involvement except for non-bulky (<7.5 cm) lymph node involvement, splenomegaly, or hepatomegaly
* Patients who have received prior antileukemic immunotherapy within 2 weeks prior to start of Isatuximab treatment
* Patients who have received treatment for leukemia with chemotherapy as follows:

Cohort 1:

* Patients who have received treatment for leukemia with chemotherapy within 2 weeks prior to start of Isatuximab treatment (exception: pre-phase therapy with 5-7 days of Dexamethasone, 3 days of Cyclophosphamide; intrathecal prophylaxis)
* Patients who are candidates for a treatment with Nelarabine

Cohort 2:

* Any chemotherapy or antibody therapy after the MRD assay leading to study inclusion (exception: intrathecal prophylaxis)
* Patients must have recovered from acute non-hematologic toxicity from previous therapies to ≤ grade I unless signs or symptoms are correlated to leukemia involvement
* Prior SCT ≤ 3 months from start of study treatment
* Acute GvHD ≥ grade II or active chronic GvHD requiring systemic treatment
* Any systemic GvHD prophylaxis or treatment within 2 weeks from start of study treatment
* Known HIV positivity, known hepatitis B surface antigen positivity or known history of hepatitis C
* Unstable or severe uncontrolled medical condition e.g. unstable cardiac function or unstable pulmonary condition
* Treatment with an investigational agent within 4 weeks from start of study treatment (safety follow-up period of respective study)
* Concurrent active malignancy other than non-melanoma skin cancer, carcinoma in situ of the cervix, or localized prostate cancer that has been treated with radiation or surgery; patients with previous malignancies are eligible if they have been disease free for ≥ 2 years and do not require any antitumor therapy.
* Evidence of uncontrolled current serious active infection or recent history (within 4 months) of deep tissue infections such as fasciitis or osteomyelitis
* Known allergies, hypersensitivity, or intolerance to boron or Mannitol, corticosteroids, mAb (including Isatuximab) or human proteins, or their excipients (refer to respective Summary of Product Characteristics), or known sensitivity to mammalian-derived products.
* Active infection, any other concurrent disease or medical condition that are deemed to interfere with the conduct of the study as judged by the investigator
* Pregnant or breastfeeding females
* Vaccination with live attenuated vaccines within 4 weeks of first study agent administration.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgement of the investigator, would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with complete hematologic response (ORR= CR and CRi) | Day 22, Week 9, per SoC
  Cohort 1:
  Proportion of patients with complete hematologic response (ORR= CR and CRi) after 2 cycles of induction therapy including Isatuximab.
Overall incidence and severity of adverse events | Day 22, Week 9, month 3, month 6 (depends on duration of therapy which is variable)
  Cohort 1:
  Overall incidence and severity of adverse events (CTCAE 5.0).
Proportion of patients with molecular response (MolCR) | Day 22, Week 9, per SoC
  Cohort 2:
  Proportion of patients with molecular response (MolCR) after one cycle of Isatuximab.

SECONDARY OUTCOMES:
Proportion of patients with CR and CRi, MolCR and cMolCR in R/R | Day 22, Week 9, per SoC
  Cohort 1:
  Proportion of patients with CR and CRi, MolCR and cMolCR in R/R (cohort 1) after 1 or 2 cycles of induction (best response)
Probability of continuous complete remission | at 18 months
  Probability of continuous complete remission (remission duration) at 18 months
Probability of overall survival | at 18 Months
  Probability of overall survival at 18 months
Probability of relapse-free survival | at 18 Months
  Probability of relapse-free survival at 18 months
Probability of event-free survival | at 18 Months
  Probability of event-free survival at 18 months
Incidence of relapses and proportion of relapse localisations | Day 22, Week 9, per SoC
  Incidence of relapses and proportion of relapse localisations
Incidence of GvHD in patients with prior SCT | until end of trial
  Incidence of GvHD in patients with prior SCT
Duration of molecular remission (mimimal residual disease by PCR) | Day 22, Week 9, per SoC
  Status is evaluated at distinct timepoints to calculate the duration of molecular remission
Treatment realization for Isatuximab | d22, week 9, per maintenance cycle, end of treatment at month 6
  Dosing of Isatuximab as scheduled per protocol
Probability of continuous MolCR and cMolCR and duration of MolCR and cMolCR | Day 22, Week 9, per SoC
  Probability of continuous MolCR and cMolCR and duration of MolCR and cMolCR
Time to MolCR and cMolCR | Day 22, Week 9, per SoC
  Time to MolCR and cMolCR measured by time-point of first achievement.
Conduct of SCT in patients with CR (ORR), MolCR, cMolCR | Through completion of the trial, average 18 months
  The conduct of SCT will be assessed in patients with CR (ORR), MolCR, cMolCR, SCT parameters and outcome
Measurement of Quality of Life | Day 22, Week 9
  Measurement of Quality of Life with EORTC instruments (e.g. EORTC QLQ-C30) at different time-points during treatment
Hospitalisation days | Day 22, Week 9, month 3 and 6 (depending on treatment duration which is individual)
  Hospitalisation days

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Goekbuget, MD, Study Director — Department of Medicine, Hematology and Oncology, Goethe University Frankfurt, Frankfurt, Germany; Anjali Cremer, MD, Principal Investigator — Department of Medicine, Hematology and Oncology, Goethe University Frankfurt, Frankfurt, Germany
Locations (14):
- Germany (14):
  - University Hospital Augsburg, II. Medizinischen Klinik, Hämatologie, internistische Onkologie und Hämostaseologie, Augsburg
  - Charité Berlin, Campus Benjamin Franklin, Department of Hematology, Oncology and Tumorimmunologyt Hämatologie, Berlin
  - Klinikum Carl Gustav Carus Dresden, Medizinische Klinik und Poliklinik I, Dresden
  - University Hospital Düsseldorf, Department of Hematology, Oncology and Clinical Immunology, Düsseldorf
  - University Hospital Erlangen AöR, Department of Medicine 5, Erlangen
  - Goethe University Hospital Frankfurt, Department of Medicine, Hematology and Oncology, Frankfurt am Main
  - University Hospital Hamburg-Eppendorf, Department of Medicine II, Hamburg
  - University Hospital Heidelberg, Department V, Hematology, Oncology and Rheumatology, Heidelberg
  - University Hospital Schleswig-Holstein, Campus Kiel, Medical Department II, Kiel
  - University Hospital Leipzig; Klinik für Hämatologie, Zelltherapie, Hämostaseologie und Infektiologie, Bereich Hämatologie und Zelltherapie, Leipzig
  - University Hospital München-Großhadern, Medizinische Klinik und Poliklinik III, München
  - University Hospital Münster, Medizinische Klinik A / KMT-Zentrum, Münster
  - Klinikum Oldenburg AöR, Universitätsklinik für Innere Medizin - Onkologie und Hämatologie, Oldenburg
  - Robert-Bosch-Krankenhaus; Abteilung für Hämatologie, Onkologie und Palliativmedizin, Stuttgart

IPD SHARING:
Plan to Share IPD: No